CLINICAL TRIAL: NCT03862495
Title: Genital Chlamydia Trachomatis Treatment to Pregnant Women to Prevent Adverse Pregnancy Outcomes: A Randomized Control Trial Pilot Study
Brief Title: Genital CT Treatment to Pregnant Women to Prevent Adverse Pregnancy Outcomes: A Pilot RCT
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-1168
Record Dates: First submitted 2019-02-22; First posted 2019-03-05 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2023-02

CONDITIONS: Chlamydia Trachomatis Infection
MeSH Terms: interventions — Azithromycin; Contact Tracing; Therapeutics

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Chlamydia Screening and Treatment (Experimental): At the time of recruitment and prior to delivery, this group will have immediate testing for C. trachomatis and N. gonorrhoeae. Physicians will notify C. trachomatis positive results to pregnant women and suggest them and their spouses to get treated according to the national standard treatment plan for Chlamydia (Azithromycin 1g, single oral administration). Patients will be followed up to confirm cure of C. trachomatis in one month. Partner notification and treatment will be suggested for pregnant women who test positive for Chlamydia.
  Interventions: Diagnostic Test: C. trachomatis and N. gonorrhoeae; Drug: Azithromycin; Other: Partner notification and treatment
- Control (Experimental): This group will have testing after delivery (immediately following childbirth) or in the event of an adverse pregnancy outcome for C. trachomatis and N. gonorrhoeae. In the event of a positive test, patients will be informed of the positive test results the same way as the intervention group. Specific treatment options will be the same as the intervention group. Physicians will ask patients to return to Nanhai Hospital one month after treatment for test of cure. Partner notification and treatment will be suggested for pregnant women who test positive for Chlamydia.
  Interventions: Diagnostic Test: C. trachomatis and N. gonorrhoeae; Drug: Azithromycin; Other: Partner notification and treatment

INTERVENTIONS:
Diagnostic Test: C. trachomatis and N. gonorrhoeae — In vitro nucleic acid amplification test for the qualitative detection of Chlamydia trachomatis and/or Neisseria gonorrhea in patient specimens utilizing amplification of target DNA by the Polymerase Chain Reaction (PCR) and nucleic acid hybridization for the detection of C. trachomatis and N. gonorrhoeae.
  Other Names: Roche Cobas Z480
Drug: Azithromycin — Azithromycin 1g administered as a single oral dose
  Other Names: Zithromax, Zmax
Other: Partner notification and treatment — Pregnant women who test positive for Chlamydia will also be suggested to take Azithromycin home to treat their spouses

SUMMARY:
This study aims to identify the relationship between genital C. trachomatis and adverse pregnancy outcomes, and investigate whether screening and treatment of genital C. trachomatis in pregnant women can reduce adverse pregnancy outcomes.

Approximately 200 pregnant women from Nanhai Hospital of Southern Medical University in Guangzhou, China will be enrolled and randomized to the intervention or control group.

DETAILED DESCRIPTION:
Women recruited for the study will be randomized to the intervention or control groups. Women in the intervention group will be tested in real time for C. trachomatis and Neisseria gonorrhoeae. Patients who test positive for either infection will be linked to physicians at the Center for treatment. For the control group, women will be tested immediately after childbirth or in the event of an adverse pregnancy outcome. In the event of a positive test result, a confirmation test will be run and if positive, the patient will be referred for treatment. The endpoint of the study is defined as either the occurrence of an adverse pregnancy outcome or delivery of a newborn.

Qualitative in-depth interviews will also be conducted with 20 of the women to explore their opinions, attitudes and feedback on the study process. University of North Carolina at Chapel Hill (UNC) investigators will work with the Nanhai Hospital of Southern Medical University and staff at Dermatology Hospital of Southern Medical University to oversee the study.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women on their first visit to the hospital (regardless of gestational age);
2. aged 18 or above;
3. agree to participate and sign an informed consent.

Exclusion Criteria:

1. systemic or topical vaginal antibiotics use within 2 weeks prior to the first perinatal visit;
2. comorbidities that are known to be related to adverse pregnancy outcomes (e.g., diabetes and hypertension);
3. diagnosed adverse pregnancy outcomes at recruitment (e.g., stillbirth); Women with a previous history of CT or NG and women with a prior adverse outcome will not be excluded. Instead, the investigators will conduct sub-analysis and check whether the intervention has different effects on different groups of pregnant women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Tang, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- China (2):
  - Dermatology Hospital of Southern Medical Hospital, Guangzhou, Guangdong
  - Nanhai Hospital of Southern Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From December 2020 to May 2023
Access Criteria: Investigator who proposes to use the data should have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chlamydia Screening and Treatment | Control
Started | 100 | 100
Completed | 63 | 65
Not Completed | 37 | 35
Not completed — Lost to Follow-up | 37 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlamydia Screening and Treatment | Control | Total
Number analyzed (Participants) | 63 | 65 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.72 (0.533) | 29.18 (0.576) | 29.45 (0.392)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 65 | 128
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 63 | 65 | 128
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 63 | 65 | 128
Premature rupture of membranes [Count of Participants; unit: Participants]
  Yes | 18 | 15 | 33
  No | 45 | 50 | 95
Premature delivery [Count of Participants; unit: Participants]
  Yes | 3 | 5 | 8
  No | 60 | 60 | 120
Low birth weight [Count of Participants; unit: Participants]
  Yes | 3 | 2 | 5
  No | 60 | 63 | 123
Pregnancy loss [Count of Participants; unit: Participants]
  Yes | 2 | 8 | 10
  No | 61 | 57 | 118

OUTCOME MEASURES:

1. Primary Outcome: Response Rate at Recruitment
Description: Number of women who get tested for CT and N. gonorrhoeae (NG) divided by the number of women being contacted about the study at the recruitment
Time Frame: at the time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Chlamydia Screening and Treatment | Control
Number analyzed (Participants) | 100 | 100
Participants | 100 | 100

2. Primary Outcome: Compliance to Receive CT or NG Treatment
Description: Number of women electing to receive CT or NG treatment within 1 week after the notification of positive test results
Time Frame: Within 1 week after the notification of positive test results
Population: Out of the 100 participants screened for each arm, 12 in the Chlamydia group tested positive and 3 in the Control group tested positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Chlamydia Screening and Treatment | Control
Number analyzed (Participants) | 12 | 3
Participants | 3 | 1

3. Primary Outcome: Number of Participants Considered as Cured After Treatment
Description: Number of women who re-tested negative either at 1 or at 3 months after treatment divided by the number of women who received CT or NG treatment
Time Frame: 1 or 3 months after the treatment
Population: Out of the 100 participants screened for each arm, 3 in the Chlamydia group were treated and 1 in the Control group was treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Chlamydia Screening and Treatment | Control
Number analyzed (Participants) | 3 | 1
Participants | 0 | 1

4. Primary Outcome: Number of Participants With Adverse Pregnancy Outcomes
Description: Number of any adverse pregnancy outcomes, including stillbirth (a baby who dies after 28 weeks of pregnancy, but before or during birth), fetal death, infant death, miscarriage (pregnancy loss between 12-28 weeks), preeclampsia (pre eclampsia: hypertension with proteinuria occurs after 20 weeks of pregnancy; eclampsia: convulsions that occur on the basis of preeclampsia and cannot be explained by other reasons), low birth weight (<2500g), smaller than gestational age, preterm birth (<37 gestational weeks), birth defect, and premature rupture of membrane (spontaneous rupture of fetal membranes before delivery, classified into full-term PROM and preterm PROM based on the gestational age) in both groups through study completion.
Time Frame: through study completion, an average of 1 year
Measure: Number; unit: participants
Arm/Group | Chlamydia Screening and Treatment | Control
Number analyzed (Participants) | 63 | 65
participants | 21 | 22

5. Secondary Outcome: Number of Participants Considered as Cured at 1 Month After the Treatment
Description: Number of women who get tested for CT and NG 1 month after the treatment divided by the number of women who receive CT or NG treatment.
Time Frame: 1 month after the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Chlamydia Screening and Treatment | Control
Number analyzed (Participants) | 63 | 65
Participants | 1 | 1

6. Secondary Outcome: Number of Participants Considered Cured at 3 Months After the Treatment
Description: Number of women who get tested for CT and NG 3 months after the treatment divided by the number of women who re-tested CT or NG positive at 1 month after the treatment
Time Frame: 3 months after the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Chlamydia Screening and Treatment | Control
Number analyzed (Participants) | 63 | 65
Participants | 1 | 1

7. Secondary Outcome: Number of People Who Completed Follow-up
Description: Number of women who are followed-up by the end of pregnancy or in the event of adverse pregnancy outcomes divided the number of women who are enrolled at the recruitment.
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Chlamydia Screening and Treatment | Control
Number analyzed (Participants) | 100 | 100
Participants | 63 | 65

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year.
Description: Given the severity of the underlying illness, participants were expected to have adverse pregnancy outcomes. All adverse pregnancy outcomes were captured as Advere Events (AEs). In addition, all Grade 3 and 4 AEs were captured as AEs in this trial. Grade 2 or higher, suspected drug-related hypersensitivity reaction was reported as an AE. All cause mortality was calculated for the ITT population, while SAEs and AEs reflect the as treated population.
Groups:
- Maternal Chlamydia Screening and Treatment: At the time of recruitment and prior to delivery, this group will have immediate testing for C. trachomatis and N. gonorrhoeae. Physicians will notify C. trachomatis positive results to pregnant women and suggest them and their spouses to get treated according to the national standard treatment plan for Chlamydia (Azithromycin 1g, single oral administration). Patients will be followed up to confirm cure of C. trachomatis in one month. Partner notification and treatment will be suggested for pregnant women who test positive for Chlamydia.
  C. trachomatis and N. gonorrhoeae: In vitro nucleic acid amplification test for the qualitative detection of Chlamydia trachomatis and/or Neisseria gonorrhea in patient specimens utilizing amplification of target DNA by the Polymerase Chain Reaction (PCR) and nucleic acid hybridization for the detection of C. trachomatis and N. gonorrhoeae.
  Azithromycin: Azithromycin 1g administered as a single oral dose
  Partner notification and treatment: Pregnant women who test positive for Chlamydia will also be suggested to take Azithromycin home to treat their spouses
- Fetus or Infant of Mother Receiving Chlamydia Screening and Treatment: Fetuses in utero or infants of mothers assigned chlamydia screening and treatment
- Maternal Control: This group will have testing after delivery (immediately following childbirth) or in the event of an adverse pregnancy outcome for C. trachomatis and N. gonorrhoeae. In the event of a positive test, patients will be informed of the positive test results the same way as the intervention group. Specific treatment options will be the same as the intervention group. Physicians will ask patients to return to Nanhai Hospital one month after treatment for test of cure. Partner notification and treatment will be suggested for pregnant women who test positive for Chlamydia.
  C. trachomatis and N. gonorrhoeae: In vitro nucleic acid amplification test for the qualitative detection of Chlamydia trachomatis and/or Neisseria gonorrhea in patient specimens utilizing amplification of target DNA by the Polymerase Chain Reaction (PCR) and nucleic acid hybridization for the detection of C. trachomatis and N. gonorrhoeae.
  Azithromycin: Azithromycin 1g administered as a single oral dose
  Partner notification and treatment: Pregnant women who test positive for Chlamydia will also be suggested to take Azithromycin home to treat their spouses
- Fetus or Infant of Mother Receiving Control: Fetuses in utero or infants of mothers assigned control
Arm/Group | Maternal Chlamydia Screening and Treatment | Fetus or Infant of Mother Receiving Chlamydia Screening and Treatment | Maternal Control | Fetus or Infant of Mother Receiving Control
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65 | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 5/65 | 21/65 | 0/63 | 22/63
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Chlamydia Screening and Treatment (N=65) | Fetus or Infant of Mother Receiving Chlamydia Screening and Treatment (N=65) | Maternal Control (N=63) | Fetus or Infant of Mother Receiving Control (N=63)
Adverse pregnancy outcomes (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 21 (26) | 0 (0) | 22 (30) — Adverse pregnancy outcomes that were also listed as the main study outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT03862495/Prot_SAP_000.pdf